CLINICAL TRIAL: NCT04977193
Title: to Evaluate the Safety and Efficacy of LY011 Cell Injection（Targeting CLDN 18.2 Chimeric Antigen Receptor T Cells） in the Treatment of Advanced Gastric Adenocarcinoma
Brief Title: A Study to Evaluate the Safety and Efficacy of ly011 Cell Injection in the Treatment of Advanced Gastric Adenocarcinoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Longyao Biotechnology Inc., Ltd. (Other)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY011C1002
Record Dates: First submitted 2021-07-12; First posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Advanced Gastric Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Biological: LY011

INTERVENTIONS:
Biological: LY011 — CAR-T

SUMMARY:
Objective to evaluate the safety and efficacy of ly011 cell injection in the treatment of advanced gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be enrolled in this study:

1. They were 18 to 70 years old, male or female; Histologically confirmed recurrent or metastatic advanced gastric adenocarcinoma (including gastric adenocarcinoma at the gastroesophageal junction);
2. Claudin 18.2 IHC staining was positive in tumor tissues;
3. Patients with advanced gastric adenocarcinoma who are not cured by second-line chemotherapy and unwilling to accept second-line chemotherapy after failure of first-line chemotherapy;
4. Life expectancy > 12 weeks;
5. According to RECIST 1.1, there was at least one measurable tumor target (≥ 10 mm);
6. ECoG scores at screening, 24 hours before puncture and baseline (before treatment) were 0-1;
7. Adequate organ function;
8. For women of childbearing age with negative pregnancy test or male subjects, effective and reliable contraceptive methods must be adopted until 30 days after the end of treatment;
9. Have enough understanding ability to voluntarily sign informed consent to participate in clinical research.

Exclusion Criteria:

Subjects who met any of the following criteria were not included in this study:

1. The patients received the following anti-tumor treatment before transplantation:

   * Cytotoxic treatment within 14 days
   * Small molecule targeted therapy for 14 days or at least 5 half lives, whichever is longer
   * Experimental drug treatment within 28 days (if the above treatment is also experimental drug treatment, the 28 day flushing period should be followed)
   * The patients were treated with monoclonal antibody within 28 days
   * Immunomodulatory therapy within 7 days
   * Radiotherapy within 14 days
2. Pregnant or lactating women;
3. Serological positive for HIV, Treponema pallidum or HCV;
4. Any uncontrollable active infection, including but not limited to active tuberculosis and HBV infection (HBsAg positive, HBcAb positive and HBV DNA positive);
5. The subjects were judged as clinically significant thyroid dysfunction by the investigators (serum thyroid hormone determination TT4, TT3, FT3, FT4, serum thyroid stimulating hormone TSH) and were not suitable to participate in this study;
6. The side effects caused by previous treatment did not recover to CTCAE ≤ 1;
7. Subjects who are currently using steroids throughout the body within 7 days before de pregnancy; Recent or recent use of inhaled steroids was not excluded;
8. Any previous treatment for claudin 18.2;
9. Previous allergy to immunotherapy and related drugs, severe allergy or allergic history;
10. T cells (including car-t and tcr-t) that have been modified by chimeric antigen receptor;
11. The subjects had untreated or symptomatic brain metastases;
12. The subjects had central or extensive lung metastases;
13. The subjects had heart disease requiring treatment or lost control of hypertension after treatment (blood pressure > 160 mmHg / 100 mmHg);
14. Subjects with a history of organ transplantation or waiting for organ transplantation;
15. There is no other serious disease that may restrict the subjects to participate in this trial;
16. The researcher assessed that the subjects were unable or unwilling to comply with the requirements of the study protocol;
17. Blood oxygen saturation ≤ 95% before treatment (receiving finger oxygen test);
18. Before pretreatment, subjects developed new arrhythmias, including but not limited to arrhythmias that could not be controlled by drugs, hypotension requiring vasopressin, bacterial, fungal or viral infections requiring intravenous antibiotics; The creatinine clearance rate was less than 40 ml / min; Investigators concluded that the subject was not suitable for further study. Subjects who use antibiotics to prevent infection can continue the trial if the researcher makes a judgment;
19. There are signs of central nervous system diseases or abnormal results of nervous system tests, which are of clinical significance;
20. The subjects were suffering from or had other malignant tumors that could not be cured within 3 years, except for cervical cancer in situ or basal cell carcinoma of skin;
21. known hypersensitivity to excipients and related adjuvants (including but not limited to dimethyl sulfoxide and dextran-40) of the study drug;
22. other conditions considered unsuitable by the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerable dose（MTD） | 1month
  MTD determination will based on the incidence of reported adverse events (including dose-limiting toxicities) and abnormal laboratory test results.
Incidence of Treatment-Emergent Adverse Events [Safety] | 2 years
  AEs according to CTCAE v 5.0.

SECONDARY OUTCOMES:
Overall Response rate（ORR） | 2 years
  the proportion of patients with best overall response of complete response (CR) or partial response (PR), as per local investigator´s assessment and according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
Area under the curve from time 0 to the last time point (AUC0-t) | 1 years
  Area under the curve from time 0 to the last time point for serum CAR-T cells
Apparent clearance (CL) | 1 years
  Apparent clearance for serum CAR-T cells
Maximum concentration (Cmax) | 1 years
  Maximum concentration for serum CAR-T cells
Half-life (T½） | 1 years
  Half-life for serum CAR-T cells
Area under the serum concentration-time curve (AUC0-inf) | 1 years
  Area under the serum concentration-time curve for serum CAR-T cells
Time to maximum concentration (Tmax) | 1 years
  Time to maximum concentration for serum CAR-T cells
Terminal elimination rate constant (λz) | 1 years
  Terminal elimination rate constant for serum CAR-T cells
Area under the curve above baseline of ANC [ANC_AUC(0-tlast)] | 1 years
  Area under the curve above baseline of ANC for serum CAR-T cells

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China